CLINICAL TRIAL: NCT00897416
Title: Validation of a Serum Marker Panel for Early Detection of Breast Cancer in High-Risk Women
Brief Title: Identification of Biomarkers in Women at High Risk or Average Risk of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Nicole Urban, ScD, Fred Hutchinson Cancer Research Center
Other Study IDs: 5518; FHCRC-5518; CDR0000355401 (Registry Identifier: PDQ)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Collecting and storing samples of blood and studying them in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is examining biomarkers in women with a high risk or average risk of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify and validate serum biomarkers that can distinguish malignant from benign and normal breast conditions in women at high risk or average risk for breast cancer.

Secondary

* Standardize procedures for recruitment, characterization, and follow-up of participants and collection, processing, storage, and analysis of specimens.
* Assess marker variability over time in healthy controls.
* Develop a shared specimen resource to support ongoing early detection research.

OUTLINE: Blood samples are collected every 6 months and assayed for the presence of biomarkers.

PROJECTED ACCRUAL: A total of 625 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Planning to undergo outpatient annual mammogram or biopsy AND meets 1 of the following criteria:

  * High risk for breast cancer
  * High risk with newly-diagnosed* breast cancer
  * Average risk for breast cancer
  * Average risk with newly-diagnosed* breast cancer
  * Benign breast disease NOTE: * Diagnosed at time of study enrollment
* No other breast cancer diagnosis within the past year
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 25 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* No hemophilia
* No other bleeding disorders

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* At least 6 months postpartum
* No planned pregnancy within the next year
* No history of medical conditions that would increase participant risk of blood draws
* No psychiatric, psychological, or other condition that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior double mastectomy

Other

* No concurrent treatment for breast cancer

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women undergoing screening mammography or breast biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 1452 (Actual)
Dates: Start 2001-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Biomarker evaluation for the early detection of breast cancer to improve outcomes for women at risk for breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Urban, ScD, Principal Investigator — Fred Hutchinson Cancer Center